CLINICAL TRIAL: NCT04004533
Title: The Development and Evaluation of a Novel Duodenoscope Assessment Tool
Status: Completed | Type: Observational
Sponsor: AdventHealth (Other)
Responsible Party: Sponsor
Other Study IDs: 1434658
Record Dates: First submitted 2019-06-05; First posted 2019-07-02 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Dudoenoscope Assessment Tool
Keywords: duodenoscope; Endoscopic retrograded cholangiopancreatography; duodenoscope assessment tool
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Endoscopic retrograde cholangiopancreatography (ERCP): At the time of each ERCP procedure, information on procedure indication, technical performance of the duodenoscope and adverse events will be collected using a newly designed duodenoscope assessment tool. The duodenoscope assessment tool was developed to measure the technical performance of the duodenoscopes based on three components: passage and positioning at the papilla, performing requisite technical maneuvers and technical features. Each performance component is graded on a scale ranging from 1 to 5 (1 for easy maneuverability, 5 for most difficult maneuverability). Duodenoscope assessment tool also captures data on procedural indications, cannulation success rates and adverse events.
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) — At the time of each ERCP procedure, information on procedure indication, technical performance of the duodenoscope and adverse events will be collected using a newly designed duodenoscope assessment tool. The duodenoscope assessment tool was developed to measure the technical performance of the duodenoscopes based on three components: passage and positioning at the papilla, performing requisite technical maneuvers and technical features. Each performance component is graded on a scale ranging from 1 to 5 (1 for easy maneuverability, 5 for most difficult maneuverability). Duodenoscope assessment tool also captures data on procedural indications, cannulation success rates and adverse events.

SUMMARY:
Endoscopic retrograde cholangiopancreatography (ERCP) procedures are performed using duodenoscopes for the treatment of pancreatic and biliary diseases. Although outcomes in endoscopic retrograde cholangiopancreatography (ERCP) procedures are measured mainly in terms of procedural success and complications, currently there are no objective tools to assess the technical performance of the duodenoscopes.

The Center for Interventional Endoscopy has maintained a multicenter database that prospectively evaluates the technical performance of duodenoscopes for performing ERCPs. Our objective is to analyze the database in order to summarize the technical performance of duodenoscopes during ERCPs and evaluate the reliability of the duodenoscope assessment tool.

DETAILED DESCRIPTION:
Outcomes in ERCP are measured mainly in terms of procedural success and complications. Recently, disposable duodenoscopes have been developed to overcome the challenges associated with reusable duodenoscope-related infections. While it is important to measure the technical performance of the newly developed disposable duodenoscope relative to conventional reusable scopes, presently, there are no objective tools to accomplish this task. The aim of this registry is to assess the reliability of a newly designed assessment tool to evaluate the technical performance of the currently available duodenoscopes. The duodenoscope assessment tool will be completed by each endoscopist after performing the ERCP and this data will be summarized and analyzed to assess the technical performance of the duodenoscopes and also to assess validity of the duodenoscope assessment tool. This is a multicenter study, with data collection from multiple centers across the United States.

ELIGIBILITY:
Inclusion Criteria

1. Aged 18 years or older
2. Undergoing ERCP using a duodenoscope

Exclusion Criteria

1. Aged less than 18 years old
2. Not undergoing ERCP using a duodenoscope

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient undergoing an ERCP with a duodenoscope and meeting the inclusion criteria will have the technical aspects of the duodenoscope function evaluated using the duodenoscope assessment tool
Sampling Method: Non-Probability Sample
Enrollment: 745 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the newly developed duodenoscope assessment tool | 6 months
  Assessment of the internal reliability of the duodenoscope assessment tool will be performed, as determined by the Cronbach's coefficient alpha

SECONDARY OUTCOMES:
Evaluation of the technical performance of duodenoscopes for performing ERCPs. | 1 day
  The technical performance of the duodenoscope during each ERCP will be based on three components: passage and positioning at the papilla, performing requisite technical maneuvers and technical features. Each performance component will be graded on a scale ranging from 1 to 5 (1 for easy maneuverability, 5 for most difficult maneuverability).
Assessment of procedural indications for ERCPs | 1 day
  The procedural indications for performing ERCPs will be assessed
Assessment of cannulation success for ERCPs | 1 day
  The number of attempts for successful cannulation of the desired duct during an ERCP will be assessed
Assessment of adverse event rates during ERCPs | 1 month
  The rate of adverse events during an ERCP will be assessed

CONTACTS AND LOCATIONS:
Overall Officials: Shyam Varadarajulu, MD, Principal Investigator — AdventHealth Orlando
Locations (9):
- United States (9):
  - University of Arkansas, Little Rock, Arkansas
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Center for Interventional Endoscopy, Orlando, Florida
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Columbia University, New York, New York
  - Allegheny Health, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Derived] Bang JY, Rosch T, Kim HM, Thakkar S, Robalino Gonzaga E, Tharian B, Inamdar S, Lee LS, Yachimski P, Jamidar P, Muniraj T, DiMaio C, Kumta N, Sethi A, Draganov P, Yang D, Seoud T, Perisetti A, Bondi G, Kirtane S, Hawes R, Wilcox CM, Kozarek R, Reddy DN, Varadarajulu S. Prospective evaluation of an assessment tool for technical performance of duodenoscopes. Dig Endosc. 2021 Jul;33(5):822-828. doi: 10.1111/den.13856. Epub 2020 Nov 17. PMID 33007136